CLINICAL TRIAL: NCT01154803
Title: Effectiveness of Nutritional Supplementation (RUTF and Multi Micronutrient) in Preventing Malnutrition in Children 6-59 Months With Infection (Malaria, Pneumonia, Diarrhoea), a Randomized Controlled Trial in Nigeria
Brief Title: Effectiveness of Nutritional Supplementation in Preventing Malnutrition in Children With Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Principal Investigator, Saskia van der Kam, Ir, Medecins Sans Frontieres, Netherlands
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MSF-nutcon02
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Malnutrition; Malaria; Lower Respiratory Tract Infection; Diarrhoea
Keywords: Supplementation; RUTF; Micronutrients; Plumpynut; Mixme; sprinkles; convalescence; weight; morbidity
MeSH Terms: conditions — Malnutrition; Malaria; Diarrhea; Convalescence; Body Weight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ready to Use Therapeutic Food (RUTF) (Experimental): 500 kcal /day for 2 weeks
  Interventions: Dietary Supplement: Ready to Use Therapeutic Food (RUTF)
- Micronutrient Powder (MNP) (Experimental): 2 x 1 g sachets micronutrients /day for 2 weeks
  Interventions: Dietary Supplement: Micronutrient Powder (MNP)
- no supplement (No Intervention): no supplementation

INTERVENTIONS:
Dietary Supplement: Ready to Use Therapeutic Food (RUTF) — 1 sachet/day, 500 kcal and multi micronutrients (fortified high quality food(RUTF),for 2 weeks after an illness (malaria, diarrhoea, pneumonia)
  Other Names: RUTF: Nutriset
  Arms: Ready to Use Therapeutic Food (RUTF)
Dietary Supplement: Micronutrient Powder (MNP) — 2 sachets / day for 14 days after an illness (diarrheoea, malaria, pneumonia)
  Other Names: MNP: DSM
  Arms: Micronutrient Powder (MNP)

SUMMARY:
The purpose of this study is to determine whether 14 days nutritional supplementation with Ready to use therapeutic Food (RUTF) or micronutrients alone to children having an infection will prevent malnutrition and reduce the frequency of morbidity.

DETAILED DESCRIPTION:
Anorexia due to infection might lead to weight loss. In many settings total recovery is problematic what might result in a permanent lower weight. A short period high quality food supplementation could improve weight gain after an infection.

A complete high quality food will be tested, but also micronutrients alone as there is no information on what children with an infection exactly need as a supplement.

Children aged 6-59 months presenting with diarrhoea, malaria or lower respiratory tract infection (LRTI) are provided for 2 weeks with

* RUTF supplement (Plumpynut®) of 500 kcal/day
* Multi-micronutrient powder (MNP)
* Placebo to MNP

The followup period is 6 months. Anthropometric indicators and morbidity are assessed monthly. Participants are invited to attend the study clinic if any signs of disease are noticed.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 59 months of age
* Not malnourished or moderately acutely malnourished children
* Diagnosis of malaria and/or diarrhoea and/or LRTI
* Intending to remain in area for the duration of the 6 month follow-up
* Living within approximately 60 minutes walking distance from the clinic
* Informed consent from a guardian*

Exclusion Criteria:

* Child is exclusively breastfeeding
* Child is severely malnourished
* Presence of 'General Danger Signs'
* Presence of severe disease (including severe malaria, severe LRTI, severe diarrhoea)
* Needing hospitalisation for any reason
* Known history of allergy to the nutritional supplementation
* Having a sibling enrolled in the study*

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2213 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
"negative nutritional outcome" of a child | 6 months follow-up
  The incidence of a negative nutritional outcome will be defined in two different ways according to the baseline nutritional status.
  i) for children with no malnourishment at time of entry into study, "negative nutritional outcome" is defined as progression to moderate or severe malnourishment ii) for children with moderate malnourishment at time of entry into study, "negative nutritional outcome" is defined as loss of ³10% of baseline weight or progression to severe malnourishment, whichever is reached first.

SECONDARY OUTCOMES:
Number of new events of a study disease | 6 months
  study disease: malaria, diarrhoea, and LRTI

CONTACTS AND LOCATIONS:
Overall Officials: Saskia Kam van der, Ir, Principal Investigator — Medecins Sans Frontieres Amsterdam
Locations (1):
- Goronyo health clinic outpatient department, Goronyo, Sokoto State, Nigeria

REFERENCES:
- [Derived] van der Kam S, Salse-Ubach N, Roll S, Swarthout T, Gayton-Toyoshima S, Jiya NM, Matsumoto A, Shanks L. Effect of Short-Term Supplementation with Ready-to-Use Therapeutic Food or Micronutrients for Children after Illness for Prevention of Malnutrition: A Randomised Controlled Trial in Nigeria. PLoS Med. 2016 Feb 9;13(2):e1001952. doi: 10.1371/journal.pmed.1001952. eCollection 2016 Feb. PMID 26859559